CLINICAL TRIAL: NCT03597282
Title: An Open-label, Phase 1B Study of NEO-PV-01 + CD40 Agonist Antibody (APX005M) or Ipilimumab With Nivolumab in Patients With Advanced or Metastatic Melanoma
Brief Title: A Personal Cancer Vaccine (NEO-PV-01) and APX005M or Ipilimumab With Nivolumab in Patients With Advanced Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed due to historically slow enrollment compounded by the COVID-19 pandemic.
Sponsor: BioNTech US Inc. (Industry)
Collaborators: Apexigen America, Inc. (Industry)
Responsible Party: Sponsor
Organization: BioNTech SE (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NT-003
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Metastatic Melanoma
Keywords: Checkpoint Inhibitor; Immunotherapy; Personalized Vaccine; Neoantigen; POLY-ICLC; Peptide
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Adjuvants, Pharmaceutic; poly ICLC; sotigalimab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- NEO-PV-01 + adjuvant + nivolumab (Experimental): Nivolumab at a dose of 240 mg will be administered by intravenous infusion (IV) every 2 weeks throughout the study. At Week 12, all patients, regardless of their disease status, will receive NEO-PV-01 + adjuvant administered subcutaneously.
  Interventions: Biological: NEO-PV-01; Biological: Nivolumab; Other: Adjuvant
- Nivolumab + adjuvant (Experimental): Nivolumab at a dose of 240 mg will be administered by intravenous infusion (IV) every 2 weeks throughout the study. At Week 12, all patients, regardless of their disease status, will receive Poly-ICLC (adjuvant) administered subcutaneously.
  Interventions: Biological: Nivolumab; Other: Adjuvant
- NEO-PV-01 + adjuvant + nivolumab on alternate schedule (Experimental): Nivolumab at a dose of 240 mg will be administered by intravenous infusion (IV) every 2 weeks throughout the study. At Week 12, all patients, regardless of their disease status, will receive NEO-PV-01 + adjuvant, administered on an alternative schedule, subcutaneously.
  Interventions: Biological: NEO-PV-01; Biological: Nivolumab; Other: Adjuvant
- NEO-PV-01 + adjuvant + nivolumab + APX005M (Experimental): Nivolumab at a dose of 240 mg will be administered by intravenous infusion (IV) every 2 weeks throughout the study. At Week 12, all patients, regardless of their disease status, will receive NEO-PV-01 + adjuvant administered subcutaneously. Patients on this arm will also receive APX005M at a dose of 0.1 mg/kg administered by IV infusion at Week 12, Week 15, and Week 19.
  Interventions: Biological: NEO-PV-01; Biological: Nivolumab; Other: Adjuvant; Biological: APX005M
- Nivolumab + APX005M (Experimental): Nivolumab at a dose of 240 mg will be administered by intravenous infusion (IV) every 2 weeks throughout the study. At Week 12, Week 15, and Week 19, all patients, regardless of their disease status, will receive APX005M at a dose of 0.1 mg/kg administered by IV infusion.
  Interventions: Biological: Nivolumab; Biological: APX005M
- NEO-PV-01 + adjuvant + nivolumab + ipilimumab (Experimental): Nivolumab at a dose of 240 mg administered by intravenous infusion (IV) every 2 weeks throughout the study. At Week 12, all patients, regardless of their disease status, will receive NEO-PV-01 + adjuvant administered subcutaneously. Patients on this arm will also receive ipilimumab at a dose of 1.0 mg/kg administered by IV infusion at Week 12 and Week 19.
  Interventions: Biological: NEO-PV-01; Biological: Nivolumab; Other: Adjuvant; Biological: ipilimumab
- Nivolumab + ipilimumab (Experimental): Nivolumab at a dose of 240 mg will be administered by intravenous infusion (IV) every 2 weeks throughout the study. At Week 12 and Week 19, all patients, regardless of their disease status, will receive ipilimumab at a dose of 1.0 mg/kg administered by IV infusion.
  Interventions: Biological: Nivolumab; Biological: ipilimumab

INTERVENTIONS:
Biological: NEO-PV-01 — Personal Cancer Vaccine
  Arms: NEO-PV-01 + adjuvant + nivolumab; NEO-PV-01 + adjuvant + nivolumab + APX005M; NEO-PV-01 + adjuvant + nivolumab + ipilimumab; NEO-PV-01 + adjuvant + nivolumab on alternate schedule
Biological: Nivolumab — monoclonal antibody against PD-1
  Other Names: Opdivo
Other: Adjuvant — immune adjuvant
  Other Names: Hiltonol; Poly-ICLC
  Arms: NEO-PV-01 + adjuvant + nivolumab; NEO-PV-01 + adjuvant + nivolumab + APX005M; NEO-PV-01 + adjuvant + nivolumab + ipilimumab; NEO-PV-01 + adjuvant + nivolumab on alternate schedule; Nivolumab + adjuvant
Biological: APX005M — monoclonal agonist antibody against CD40
  Arms: NEO-PV-01 + adjuvant + nivolumab + APX005M; Nivolumab + APX005M
Biological: ipilimumab — monoclonal antibody against CTLA4
  Other Names: Yervoy
  Arms: NEO-PV-01 + adjuvant + nivolumab + ipilimumab; Nivolumab + ipilimumab

SUMMARY:
The primary purpose of this study is to demonstrate that the NEO-PV-01 vaccine, either with APX005M or ipilimumab, and nivolumab is safe for the treatment of patients with advanced or metastatic melanoma. The study will also investigate an alternative schedule for the administration of the NEO-PV-01 vaccine. Study interventions will be assessed by both clinical and immune responses to treatment.

DETAILED DESCRIPTION:
This clinical trial will enroll patients with advanced or metastatic melanoma not having received treatment for metastatic disease. The 5 agents being used in this study are:

* A new, investigational, personal cancer vaccine called "NEO-PV-01".
* Poly-ICLC (Hiltonol), an investigational adjuvant that is used to help stimulate the immune system.
* A cancer drug called APX005M, a drug that stimulates specific types of immune cells that help the immune system to recognize specific targets.
* A cancer drug called ipilimumab
* A cancer drug called nivolumab

NEO-PV-01, APX005M, ipilimumab, and nivolumab are considered immunotherapies and work using the immune system to fight cancer. NEO-PV-01 is a personal vaccine therapy in that it is manufactured specifically to include targets for the immune system that are present uniquely on your cancer. Poly-ICLC is an adjuvant that helps stimulate the immune system and make the vaccine, NEO-PV-01, more effective.

The purpose of this study is to find out if treatment with NEO-PV-01 + Poly-ICLC (the NEO-PV-01 vaccine) in combination with either APX005M or ipilimumab, and nivolumab is safe and useful for patients with melanoma. The study also will assess if the NEO-PV-01 vaccine, when given at different intervals, can improve your response compared with the standard schedule. This study will also assess the effects of poly-ICLC in combination with nivolumab. The side effects of all study drugs will be monitored and additional research tests will be done to assess your immune response to your cancer. There is no guarantee that you will benefit from therapy with the study drugs.

The FDA has not yet approved the NEO-PV-01 vaccine for use alone or in combination with other cancer drugs such as APX005M, ipilimumab, and nivolumab. Neither APX005M nor Poly-ICLC are approved for use in your type of cancer. Ipilimumab and nivolumab are both approved for use in your type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent.
* Age ≥ 18 years.
* Have cytologically or histologically confirmed advanced or metastatic melanoma and having received no prior systemic therapy for metastatic disease.
* Have at least 1 site of disease measurable by RECIST 1.1 that has not been treated with local therapy within 6 months of study treatment. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Have at least 1 site of disease accessible to repeat biopsies for tumor sequencing and immunological analysis. This site may be a target lesion as long as it will not become unmeasurable by the biopsy procedure.
* Have Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1 with an anticipated life expectancy of > 6 months.
* Recovered from all toxicities associated with prior treatment to acceptable baseline status (for laboratory toxicities, see below limits for inclusion) or a National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03, Grade of 0 or 1, except for toxicities not considered a safety risk (e.g., alopecia or vitiligo).
* Screening laboratory values must meet the following criteria and should be obtained within 30 days (or 45 days if a biopsy is repeated) prior to study treatment:

  1. White blood cell (WBC) count ≥ 3 × 103/µL
  2. Platelet count ≥ 100 × 103/µL
  3. Hemoglobin > 9 g/dL
  4. Serum creatinine ≤ 1.5 × upper limit of normal (ULN)
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN or ≤ 5 × ULN for patients with liver metastases
  6. Total bilirubin ≤ 1.5 × ULN (except in patients with Gilbert Syndrome who can have total bilirubin < 3.0 mg/dL).
* Female patients of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female patients of childbearing potential must be willing to use an adequate method of contraception, as outlined in the protocol, for the course of the study through 120 days after last dose of study medication.
* Male patients of childbearing potential must agree to use an adequate method of contraception, as outlined in the protocol, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

Exclusion Criteria

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of first dose of treatment.
* Received any systemic therapy for advanced or metastatic cancer treatment including immunotherapeutic agents such as anti-programmed cell death protein 1 (anti-PD-1), anti-PD-L1, anti-CD40, or anti-cytotoxic T-lymphocyte-associated antigen 4 (anti-CTLA-4) antibody therapy.
* Have had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from AE due to agents administered more than 4 weeks earlier.
* Have had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 30 days prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from AEs due to a previously administered agent.

  1. Note: Patients with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study.
  2. Note: If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Received radiation therapy at the biopsy sites.
* Received prior tyrosine kinase inhibitor therapy or palliative radiation within 7 days of Cycle 1/Day 1.
* Have known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging [using the identical imaging modality for each assessment, either magnetic resonance imaging (MRI) or computed tomography (CT) scan] for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Have active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Have a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
* Received a live vaccination within 30 days of planned treatment start date.
* Have an active infection requiring systemic therapy.
* Have a history of sensitivity or allergy to mAbs or immunoglobulin G (IgG).
* Have a history of allogeneic bone marrow transplantation.
* Have a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Have known active Hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or Hepatitis C (e.g., hepatitis C virus [HCV] RNA [qualitative] is detected).
* Have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring treatment, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
* Have any underlying medical condition, psychiatric condition, or social situation that, in the opinion of the Investigator, would compromise study administration as per protocol or compromise the assessment of AEs.
* Have a planned major surgery.
* Are pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Nursing women are excluded from this study because there is an unknown but potential risk of AEs in nursing infants secondary to treatment of the mother with nivolumab, personalized neoantigen peptides, adjuvant, ipilimumab, and APX005M.
* Have a history of additional invasive metastatic disease (other than melanoma), except for the following:

  1. Individuals with a history of invasive metastatic disease are eligible if they have been disease free for at least 2 years and are deemed by the Investigator to be at low risk for recurrence of that metastatic disease;
  2. Individuals with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or local papillary thyroid cancer, who have undergone therapy with curative intent.
* Have severe hypersensitivity (≥ Grade 3) to nivolumab and/or any of its excipients.
* Have mucosal melanoma, uveal melanoma, or acral lentiginous melanoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
The rate of adverse events and severe adverse events leading to treatment discontinuation | Baseline through 90 days after the last dose of nivolumab
  Rate of adverse events and severe adverse events leading to treatment discontinuation and those adverse events and severe adverse events detected during symptom-directed physical examinations (changes in safety laboratory evaluations, physical examination findings. vital signs, and ECOG PS)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline through 52 weeks
  Objective Response Rate (ORR), defined as the proportion of patients who achieve complete response (CR) or partial response (PR) based on Response Criteria in Solid Tumors (RECIST) v1.1
Clinical Benefit Rate | Baseline through 52 weeks
  Clinical Benefit Rate (CBR), defined as the proportion of patients who achieve a CR, PR, or stable disease (SD) based on RECIST v1.1
Duration of response | Baseline through 52 weeks
  Duration of Response (DOR) defined as the date of the first documentation of a confirmed response to the date of the first documented progressive disease (PD) based on RECIST v1.1
Response conversion rate | Baseline through 52 weeks
  Response Conversion Rate (RCR), defined as the proportion of patients who improve in RECIST v1.1 category subsequent to vaccination (eg. PD to SD/PR/CR, SD to PR/CR, PR to CR).
Progression free survival | Baseline through 52 weeks
  Progression Free Survival (PFS), defined as the time from the date of first dosing to the date of first documented PD or death
Overall survival | Baseline through up to 3 years
  Overall Survival (OS), defined from the date of enrollment and death from any cause

OTHER OUTCOMES:
Immune Responses | Baseline through 52 weeks
  Antigen-specificity in peripheral CD8+ and CD4+ T cell responses and biomarker analyses of tumor biopsies following treatment
Overall response rate | Baseline through 52 weeks
  To determine the anti-tumor activity, as assessed by ORR by iRECIST
Progression free survival | Baseline through 52 weeks
  To determine the anti-tumor activity, as assessed by PFS by iRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Mark DeMario, MD, Study Director — BioNTech US Inc.
Locations (8):
- United States (8):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - University of Colorado Denver, Denver, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No